CLINICAL TRIAL: NCT01288872
Title: Praziquantel Pharmacokinetics in Pregnancy and During Lactation
Brief Title: Praziquantel-Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-0049; 5U01AI066050-07 (NIH)
Record Dates: First submitted 2011-01-28; First posted 2011-02-03 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2013-09

CONDITIONS: Schistosomiasis
Keywords: Praziquantal, Schistosomiasis, pregnant women, Philippines
MeSH Terms: conditions — Schistosomiasis | interventions — Praziquantel

ARMS (1):
- Praziquantel (Experimental): 45 women in 3 cohorts (15 early pregnancy: 12-16 weeks gestation; 15 late pregnancy: 30-36 weeks gestation; and 15 lactating nonpregnant women who are 5-7 months (inclusive) postpartum) given praziquantel (PZQ), 60 mg/kg orally in split dose (30 mg/kg each) separated by 3 hours.
  Interventions: Drug: Praziquantel

INTERVENTIONS:
Drug: Praziquantel — Praziquantel (PZQ), 60 mg/kg, administered orally in split dose (30 mg/kg each dose) separated by three hours.

SUMMARY:
The purpose of the study is to understand whether the drug praziquantel (PZQ) is metabolized or broken down differently when women are pregnant versus not pregnant. PZQ is used to treat schistosomiasis (worm infection). Researchers will study how PZQ is broken down among 15 women who are 12-16 weeks pregnant, 15 women who are 30-36 weeks pregnant, and 15 women nonpregnant women who are producing breast milk. All women will be 18 or older and otherwise healthy. The usual practice is to wait until after mothers have finished pregnancy and breast feeding before giving PZQ. Participants will receive 2 doses of PZQ separated by 3 hours. Study procedures will include a 24 hour hospital stay following administration of PZQ, blood, stool and urine samples, ultrasound if pregnant, and physical exams of mother and baby. Patient participation for mother/infant pair is about 9 months.

DETAILED DESCRIPTION:
Schistosomiasis infects over 200 million individuals and remains a significant cause of morbidity and mortality in developing countries, despite the availability of effective pharmacologic therapy with praziquantel (PZQ). Researchers propose to conduct a phase I study of the pharmacokinetics (PK) and safety of PZQ for the treatment of Schistosomiasis (S.) japonicum among pregnant and lactating women living in the province of Leyte, The Philippines. In practice, treatment of schistosomiasis is withheld for both pregnant and lactating post partum women in the Philippines as well as other countries endemic for schistosomiasis. Without treatment, these women accrue known morbidities identified among non-pregnant subjects including hepatic fibrosis, under-nutrition, and anemia. The overall aims of this study are to see if there are differences in PZQ PK and safety during pregnancy compared to post partum, to describe the kinetics of breast milk transfer of PZQ and to estimate the dose of PZQ received by a nursing infant whose mother is treated with PZQ. This protocol will enroll 15 pregnant women in early pregnancy (12-16 weeks gestation), 15 pregnant women in late pregnancy (30-36 weeks gestation) and 15 lactating nonpregnant women between 5 and 7 months postpartum. The study population will consist of S. japonicum infected women in study villages or at the Municipal Health Centers. Women must be: age 18 or older, otherwise healthy without disease of any major organ system, without history of seizures, chronic medical problem or any neurologic disorders, without history of severe allergic reaction to PZQ and willing to provide informed consent to participate. The pregnant women must: have a singleton pregnancy, be carrying a fetus without evidence of anomaly by ultrasound. Pregnant subjects will be treated with PZQ in early pregnancy (12-16 weeks gestation) or late pregnancy (30-36 weeks gestation), lactating nonpregnant (5-7 months postpartum inclusive ). A total dose of 60 mg/kg of study medication will be provided in 2 split doses over 3 hours as this has been shown to substantially reduce drug side effects. All subjects will be hospitalized overnight for intensive blood sampling and for monitoring for adverse events. Serial breast milk samples will be collected from lactating women. Plasma and breast milk will be assayed for PZQ concentration. PK parameters in pregnant and postpartum women will be compared and kinetics of praziquantel breast milk transfer and estimation of infant PZQ dose from breast milk will be determined. Safety assessments will be performed on pregnant women and their infants through 1 month postpartum, and on postpartum women through 2 weeks post dosing. This study is linked to Division of Microbiology and Infectious Disease (DMID) protocol 06-0039.

ELIGIBILITY:
Inclusion Criteria:

Screening:

* Woman must be age 18 or over.
* Present to a study midwife or health center.
* Live in a study village.

Inclusion criteria for the study are as follows:

* Infected with Schistosomiasis (S.) japonicum.
* Age 18 or older.
* Participant is otherwise healthy as determined by history, physical exam, ultrasound (if pregnant) and laboratory assessment, with the exception of laboratory values cited in Exclusion Criteria.
* Early pregnancy cohort: pregnant, between 12-16 weeks gestation.
* Late pregnancy cohort: pregnant, between 30-36 weeks gestation
* Lactating nonpregnant: 5-7 months postpartum inclusive (up to 7 months and 31 days) with negative pregnancy test.
* Ability to provide informed consent to participate.

Exclusion Criteria:

* Presence of significant disease/illness that is either acute or chronic. This will be defined by history, physical examination, ultrasound (if pregnant) and laboratory assessment. In particular:

  1. History of seizures or other neurologic disorder, chronic medical problem determined by history or physical examination, e.g., active hepatitis, renal disease, tuberculosis, heart disease.
  2. Grade 3 or higher laboratory abnormality of blood urea nitrogen (BUN), creatinine, bilirubin, white blood cell count, or platelet count will warrant exclusion. Grade 2 or higher abnormality of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) will warrant exclusion. For hemoglobin, women with severe anemia defined as hemoglobin less than 7.0 g/dL will be excluded.
  3. If pregnant, with myoma on ultrasound that are sub-mucosal OR women with myoma that are in any location and greater than 5 cm in size.
  4. If pregnant, with congenital anomalies of the reproductive tract that would be expected to cause decreased fetal weight or greatly increase the risk of pre-maturity such as duplicate uterus, uterine septum.
  5. For less clear cases, we will define significant illness as one that significantly alters a woman's ability to perform activities of daily living, causes symptoms at least two days per week, or necessitates regular use of medication. In the case of acute medical conditions, such as urinary tract infection, pneumonia, or febrile illness, enrollment may be postponed until the illness is successfully treated (not currently on any medication for the illness).
* For lactating postpartum subjects: milk supply suspected to be marginal so that 24 hour interruption of nursing likely to lead to inability to restart breast feeding, evidence of breast infection, or history of breast surgery.
* Presence of cysts in the eye suggestive of neurocysticercosis.
* Regular use of a medication for a chronic medical condition.
* History of severe allergic reaction (anaphylaxis, facial swelling, or difficulty breathing) or seizure with praziquantel administration.
* If pregnant, fetus has congenital anomaly determined by ultrasound or is determined to be nonviable e.g., blighted ovum.
* Twin or higher order pregnancy.
* Woman has been enrolled into this study or its companion study ("S. japonicum and pregnancy outcomes: A Randomized, Double Blind, Placebo Controlled Trial (RCT). DMID Protocol Number: 06-0039") for a previous pregnancy.
* Inability to comprehend study procedures and provide informed consent due to limited cognitive abilities or other reason, or refuses to provide informed consent.
* Subjects receiving during the previous month any of the following drugs which may interact with praziquantel (PZQ) bioavailability, metabolism and/or elimination: carbamazepine, chloroquine, cimetidine, dexamethasone, erythromycin, fosphenytoin, itraconazole, ketoconazole, phenobarbital, phenytoin, rifampin, or any protease inhibitor or non-nucleoside reverse transcriptase inhibitor.
* Subjects ingesting grapefruit juice during the previous week.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Comparison of PZQ and 4-hydroxy PZQ PK parameters in pregnant and nonpregnant lactating subjects, central tendency and distribution (Cmax, Tmax, t ½, AUC, CL/F and Vd/F). | Up to 24 hours after the first dose of PZQ
Early Pregnancy Cohort only: Assessed for the presence of pre-eclampsia. | Assessed for the presence of pre-eclampsia at both the 22 and 32 week visits.
Pregnant women only: newborn congenital anomalies. The number of infants with congenital anomalies | Newborn examined by the midwife (or pediatrician if in hospital) at delivery and within 2-6 days of delivery to assess the presence of congenital anomalies and well-being. Newborn examined by study pediatrician at 28 days of life.
Early Pregnancy Cohort only: number of subjects experiencing a spontaneous abortion and number of stillbirths reported after drug administration; and live birth rate among pregnant subjects. | Women will be observed in hospital for 24 hours after dosing and asked to return for any bleeding at any time.
Toxicity to maternal bone marrow, kidney, and liver will be assessed by measurement of complete blood count, blood urea nitrogen (BUN) and creatinine, and liver function tests (AST, ALT, and bilirubin). | Collected just before the dose, 24 hours after the dose and at either 20 weeks after the dose (early gestation subjects) or 10-14 days after the dose (late gestation and lactating postpartum subjects).
Subjects will be observed in hospital for adverse events/serious adverse events (AE/SAEs). | Up to 9 months from enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute for Tropical Medicine - Health Compound, Muntinlupa City, National Capital Region, Philippines